CLINICAL TRIAL: NCT01220752
Title: Treatment of Malignant Sinonasal Tumours With Intensity-modulated Radiotherapy (IMRT) and Carbon Ion Boost (C12)
Acronym: IMRT-HIT-SNT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Alexandra Jensen, Investigator, Heidelberg University
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IMRT-HIT-SNT
Record Dates: First submitted 2010-10-12; First posted 2010-10-14 (Estimated); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Sinonasal Malignancies; Adenocarcinoma and Squamous Cell Carcinoma of the Paranasal Sinuses
Keywords: IMRT; carbon ion therapy; paranasal sinus; nasal cavity; adenocarcinoma; squamous cell carcinoma
MeSH Terms: conditions — Adenocarcinoma; Carcinoma, Squamous Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMRT + carbon ion boost (Experimental): (8 x 3 GyE) carbon ion therapy followed by 50 Gy IMRT (2 Gy/ Fx)corresponding to a total dose of approximately 74 GyE.
  Interventions: Radiation: carbon ion boost

INTERVENTIONS:
Radiation: carbon ion boost — 8 fractions carbon ion (8 x 3 GyE C12) therapy followed by 25 fractions of IMRT corresponding to a total dose of approximately 74 GyE. Treatment duration is approximately 61/2-7 weeks

SUMMARY:
The IMRT-HIT-SNT trial is a prospective, mono-centric, phase II trial evaluating toxicity and efficacy in the combined treatment with intensity-modulated radiation therapy (IMRT) and carbon ion (C12) boost. Primary endpoint is mucositis ≥ CTC°3, secondary endpoints are local control, disease-free survival, overall survival, and toxicity. Planned accrual of the trial includes 36 patients with histologically proven (≥R1-resected or inoperable) sinonasal malignancies.

DETAILED DESCRIPTION:
Local control in sinonasal malignancies is dose dependent. However, dose escalation at acceptable toxicity is technically demanding even with modern radiotherapy techniques. Raster-scanned carbon ion therapy with highly conformal dose distributions may allow higher doses at comparable or reduced side-effects.

Methods/ design:

The IMRT-HIT-SNT trial is a prospective, mono-centric, phase II trial evaluating toxicity in the combined treatment with intensity-modulated radiation therapy (IMRT) and carbon ion (C12) boost in 36 patients with histologically proven (≥R1-resected or inoperable) adeno-/ or squamous cell carcinoma of the nasal cavity or paransal sinuses. Patients receive 24 GyE carbon ions (8 fractions) and IMRT (2.0 Gy/ fraction).

Study objectives:

Incidence of mucositis ≥ CTC°3 will be assessed as the primary endpoint of the trial, local control, disease-free survival, overall survival, and toxicity (incl. mucositis CTC °I-II and late toxicity at 2 years post RT)are secondary endpoints.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed or surgically removed adenocarcinoma or squamous cell carcinoma of the nasal cavity or paranasal sinuses
* Inoperable tumour or refusal to undergo surgical resection
* Macroscopic or microscopic residual tumour (R2/ R1) or
* ≥T3/T4 or
* written informed consent
* pts aged 18 - 80 years
* effective contraception for pts in childbearing age (<12 months post beginning of menopause)

Exclusion Criteria:

* Prior radio- or chemotherapy for tumours of the head and neck
* Other previous malignancy within the past 5 years except prior, adequately treated basal cell carcinoma of the skin or pre-invasive carcinoma of the cervix
* Significant neurological or psychiatric condition including dementia or seizures or other serious medical condition prohibiting the patient's participation in the trial by judgement of the investigators
* Legal incapacity or limited legal capacity
* Positive serum/ urine beta-HCG/ pregnancy
* Drug abuse

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06-17 (Actual); Primary Completion 2019-08-29 (Actual); Study Completion 2021-12-19 (Actual)

PRIMARY OUTCOMES:
mucositis CTC grade 3 | 6-8 weeks post completion of treatment
  Incidence of mucositis ≥ CTC°III will be assessed as the primary endpoint of the trial at completion of radiation therapy

SECONDARY OUTCOMES:
local control | 2 years post completion of RT
disease-free survival | 2 years post completion of RT
overall survival | 2 years post completion of RT
acute toxicity CTC grade 1/2 | within 90 days of RT
late toxicity | from 90 days to trial completion

CONTACTS AND LOCATIONS:
Overall Officials: Juergen Debus, MD PhD, Principal Investigator — Heidelberg University
Locations (1):
- Dept of Radiation Oncology, University of Heidelberg, INF 400, Heidelberg, Germany

REFERENCES:
- [Background] Muir CS, Nectoux J. Descriptive epidemiology of malignant neoplasms of nose, nasal cavities, middle ear and accessory sinuses. Clin Otolaryngol Allied Sci. 1980 Jun;5(3):195-211. doi: 10.1111/j.1365-2273.1980.tb01647.x. PMID 6996871
- [Background] Roush GC. Epidemiology of cancer of the nose and paranasal sinuses: current concepts. Head Neck Surg. 1979 Sep-Oct;2(1):3-11. doi: 10.1002/hed.2890020103. PMID 400658
- [Background] Madani I, Bonte K, Vakaet L, Boterberg T, De Neve W. Intensity-modulated radiotherapy for sinonasal tumors: Ghent University Hospital update. Int J Radiat Oncol Biol Phys. 2009 Feb 1;73(2):424-32. doi: 10.1016/j.ijrobp.2008.04.037. Epub 2008 Aug 26. PMID 18755554
- [Background] Licitra L, Locati LD, Cavina R, Garassino I, Mattavelli F, Pizzi N, Quattrone P, Valagussa P, Gianni L, Bonadonna G, Solero CL, Cantu G. Primary chemotherapy followed by anterior craniofacial resection and radiotherapy for paranasal cancer. Ann Oncol. 2003 Mar;14(3):367-72. doi: 10.1093/annonc/mdg113. PMID 12598339
- [Background] Dulguerov P, Jacobsen MS, Allal AS, Lehmann W, Calcaterra T. Nasal and paranasal sinus carcinoma: are we making progress? A series of 220 patients and a systematic review. Cancer. 2001 Dec 15;92(12):3012-29. doi: 10.1002/1097-0142(20011215)92:123.0.co;2-e. PMID 11753979
- [Background] Parsons JT, Mendenhall WM, Mancuso AA, Cassisi NJ, Million RR. Malignant tumors of the nasal cavity and ethmoid and sphenoid sinuses. Int J Radiat Oncol Biol Phys. 1988 Jan;14(1):11-22. doi: 10.1016/0360-3016(88)90044-2. PMID 3335447
- [Background] Shukovsky LJ, Fletcher GH. Retinal and optic nerve complications in a high dose irradiation technique of ethmoid sinus and nasal cavity. Radiology. 1972 Sep;104(3):629-34. doi: 10.1148/104.3.629. No abstract available. PMID 4626287
- [Background] Brizel DM, Light K, Zhou SM, Marks LB. Conformal radiation therapy treatment planning reduces the dose to the optic structures for patients with tumors of the paranasal sinuses. Radiother Oncol. 1999 Jun;51(3):215-8. doi: 10.1016/s0167-8140(99)00043-2. PMID 10435816
- [Background] Huang D, Xia P, Akazawa P, Akazawa C, Quivey JM, Verhey LJ, Kaplan M, Lee N. Comparison of treatment plans using intensity-modulated radiotherapy and three-dimensional conformal radiotherapy for paranasal sinus carcinoma. Int J Radiat Oncol Biol Phys. 2003 May 1;56(1):158-68. doi: 10.1016/s0360-3016(03)00080-4. PMID 12694834
- [Background] Lomax AJ, Goitein M, Adams J. Intensity modulation in radiotherapy: photons versus protons in the paranasal sinus. Radiother Oncol. 2003 Jan;66(1):11-8. doi: 10.1016/s0167-8140(02)00308-0. PMID 12559516
- [Background] Mock U, Georg D, Bogner J, Auberger T, Potter R. Treatment planning comparison of conventional, 3D conformal, and intensity-modulated photon (IMRT) and proton therapy for paranasal sinus carcinoma. Int J Radiat Oncol Biol Phys. 2004 Jan 1;58(1):147-54. doi: 10.1016/s0360-3016(03)01452-4. PMID 14697432
- [Background] Hoppe BS, Wolden SL, Zelefsky MJ, Mechalakos JG, Shah JP, Kraus DH, Lee N. Postoperative intensity-modulated radiation therapy for cancers of the paranasal sinuses, nasal cavity, and lacrimal glands: technique, early outcomes, and toxicity. Head Neck. 2008 Jul;30(7):925-32. doi: 10.1002/hed.20800. PMID 18302261
- [Background] Truong MT, Kamat UR, Liebsch NJ, Curry WT, Lin DT, Barker FG 2nd, Loeffler JS, Chan AW. Proton radiation therapy for primary sphenoid sinus malignancies: treatment outcome and prognostic factors. Head Neck. 2009 Oct;31(10):1297-308. doi: 10.1002/hed.21092. PMID 19536762
- [Background] Hoppe BS, Nelson CJ, Gomez DR, Stegman LD, Wu AJ, Wolden SL, Pfister DG, Zelefsky MJ, Shah JP, Kraus DH, Lee NY. Unresectable carcinoma of the paranasal sinuses: outcomes and toxicities. Int J Radiat Oncol Biol Phys. 2008 Nov 1;72(3):763-9. doi: 10.1016/j.ijrobp.2008.01.038. Epub 2008 Apr 18. PMID 18395361
- [Background] Therasse P, Arbuck SG, Eisenhauer EA, Wanders J, Kaplan RS, Rubinstein L, Verweij J, Van Glabbeke M, van Oosterom AT, Christian MC, Gwyther SG. New guidelines to evaluate the response to treatment in solid tumors. European Organization for Research and Treatment of Cancer, National Cancer Institute of the United States, National Cancer Institute of Canada. J Natl Cancer Inst. 2000 Feb 2;92(3):205-16. doi: 10.1093/jnci/92.3.205. PMID 10655437
- [Derived] Jensen AD, Nikoghosyan AV, Windemuth-Kieselbach C, Debus J, Munter MW. Treatment of malignant sinonasal tumours with intensity-modulated radiotherapy (IMRT) and carbon ion boost (C12). BMC Cancer. 2011 May 22;11:190. doi: 10.1186/1471-2407-11-190. PMID 21600049